CLINICAL TRIAL: NCT04334434
Title: Investigation Of The Effectiveness Of The Telerehabilitation Applied To Individuals Over The Age Of 65 Who Experience Social Isolation At Houses Due To The Coronavirus (Covid-19) Pandemic
Brief Title: Telerehabilitation in Individuals Over 65 Years of Age Having Social Isolation Due to Coronavirus (Covid-19)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kubra Koce, MSc PT (Other)
Responsible Party: Sponsor-Investigator, Kubra Koce, MSc PT, Physiotherapist, MSc, Istanbul University - Cerrahpasa
Organization: Istanbul University - Cerrahpasa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 002
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Telerehabilitation
Keywords: Covid-19; Exercises; Social Isolation
MeSH Terms: conditions — COVID-19; Motor Activity; Social Isolation | interventions — Telerehabilitation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): The group to which the exercise protocol consisting of aerobic and strengthening exercises will be applied.
  Interventions: Other: Telerehabilitation
- Control Group (No Intervention): Control group where evaluations will be made.

INTERVENTIONS:
Other: Telerehabilitation — 15 volunteers over 65 years old who are at home during the social isolation process due to the coronavirus outbreak will be included in this group. An online exercise protocol was created for individuals who will participate in the study. Each exercise session was planned as 30 minutes for 3 days a week for 4 weeks. It was planned to start the protocol with warm-up exercises and finish with cooling exercises. The exercise protocol was additionally determined as a combination of aerobic and strengthening exercises. Individuals were asked to participate in the study via Skype and aimed to do their exercises with a physiotherapist
  Arms: Study Group

SUMMARY:
In December 2019, new coronavirus pneumonia (COVID-19) erupted in Wuhan (Hubei, China) and quickly spread from a single city to the entire country in just 30 days and then attracted worldwide attention. COVID-19 causes a large number of deaths due to its occurrence in many cases. This virus caused a total of 549,461 approved cases and 24,887 deaths worldwide. All the countries of the world take some precautions to prevent the spread of this epidemic disease, which WHO declared it as "pandemic". Staying home and social isolation are at the top of these precautions. For this purpose, in Turkey on March 21, 2020, '65 and older individuals began to apply the curfew to individuals with chronic illnesses. However, not leaving the house and social isolation brings with it the limitation of physical activity. Physical activity (PA) is defined by WHO as any bodily movement produced by the contraction of skeletal muscles that increases energy consumption. Recommended PA levels for the elderly (≥65 years) are similar to adults (18 to 64 years old). At the global level, approximately 45% of people over the age of 60 do not meet the recommended level of PA. Studies investigating the relationship between social isolation and health behavior report consistent findings. Individuals with smaller social networks report less healthy diets, excessive alcohol consumption, and less physical activity. The effects of social isolation are related to physical inactivity, smoking and the possibility of having both health risk behaviors together. The decrease in physical performance is associated with the risk of falling, sarcopenia, fragility, decreased quality of life, emotionalization, comorbidity, early death, and increased health care costs. Practical and innovative interventions are needed to reduce the decline in muscle mass, strength and physical performance in the aging population. When today's conditions are evaluated, technology-supported education programs are effective in increasing the motivation for physical activity. The purpose of this study; to evaluate the physical activity level of individuals over the age of 65 who experience social isolation due to the precautions taken in our country to prevent the spread of the COVID-19 pandemic, and to investigate the effectiveness of home-based telerehabilitation exercises. It is aimed to use an innovative model based on the digitally supported, home-based exercise program.

ELIGIBILITY:
Inclusion Criteria:

* Being 65 years old and over
* Being in social isolation due to the coronavirus epidemic.
* Spending at least 1 week at home different from routine life.
* Not to be obstructed from doing physical activities.
* To have access to online exercise training.

Exclusion Criteria:

* Having a serious cognitive impairment
* Having serious hearing and vision problems
* Having vestibular disorders that can cause loss of balance
* Having diabetes, hypertension or a neurological disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Physical Activity Scale for the Elderly | 2 weeks
  One of the evaluation parameters created to evaluate the physical activity level of elderly individuals, the factors affecting the activity level, the relationship between physical activity and health profile is the Physical Activity Scale for the Elderly. The minimum score that can be obtained from the scale is 0 and the maximum score is 400. The higher score on the scale indicates a better level of physical activity.
Nottingham Health Profile | 2 weeks
  Nottingham Health Profile was created in England in 1985 to evaluate the quality of life-related to health. The Nottingham Health Profile is a general quality of life questionnaire that assesses the level of individuals health problems and how they affect their daily life activities.
Loneliness Scale for the Elderly | 2 weeks.
  It was created by Gierveld and Kamphuis in 1985 to evaluate the sense of loneliness in older individuals and was revised in 1999 by Tilburg and Gierveld. It consists of 11 items in total and two subtitles.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul university Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No